CLINICAL TRIAL: NCT01250964
Title: Endothelial Cell Loss and Surgically Induced Astigmatism After 2.2 mm Wound Assisted vs 2.4 mm Wound-Directed Clear Corneal Incisions for Intraocular Lens Insertion During Cataract Surgery
Brief Title: Endothelial Cell Loss and Induced Astigmatism After Wound-directed and Wound-assisted IOL Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Dr. Kenneth Cohen, Dept. of Ophthalmology, UNC Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0435
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Cataracts; Cataract Surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound-assisted lens injection (Active Comparator): Wound-assisted lens injection is considered neither superior or inferior to wound-directed lens injection.
  Interventions: Procedure: Lens insertion during cataract surgery
- Wound-directed lens injection (Active Comparator): Wound-directed lens injection is neither considered superior nor inferior to wound-assisted lens injection.
  Interventions: Procedure: Lens insertion during cataract surgery

INTERVENTIONS:
Procedure: Lens insertion during cataract surgery — After cataract removal during cataract surgery, a lens needs to be injected into the eye. Both arms are routinely used but different methods for injecting the lens.

SUMMARY:
The purpose of this study is to determine if there is any difference in astigmatism (eye surface curvature) or corneal endothelial cell density (the inner cell lining of the eye surface) after two different methods for inserting a lens during cataract surgery.

DETAILED DESCRIPTION:
Cataract surgery (removal of a cloudy lens) is currently performed through increasingly smaller incisions. Bimanual surgery, where two instruments are used to remove the lens, is performed through two 1.4 mm incisions. Typically, one of these incisions is enlarged to 2.2 or 2.4 mm in order that the IOL (artificial lens) can be inserted into the eye. Surgeons insert these lenses by placing a lens injector cartridge completely into the eye (wound-directed insertion) or by placing only the tip inside the incision (wound-assisted insertion). While wound-assisted insertion can be performed through slightly smaller incisions (2.2 mm versus 2.4 mm for wound-directed insertion), both methods of insertion cause some incision enlargement. There is some evidence that wound-assisted insertion can cause very short-term pressure within the eye to go up. Neither method is considered inferior or superior to the other, and the primary investigator (Dr. Kenneth Cohen) routinely uses both methods.

No studies have directly compared wound-healing characteristics between these two methods. We seek to compare differences in:

1. Surgically-induced astigmatism (changes in the corneal curvature from cataract surgery incisions.
2. Endothelial cell density loss. Endothelial cells line the inside surface of the cornea, and their overall density can be decreased by cataract surgery.
3. Best-corrected vision after surgery
4. Sizes of the incisions after lens injection

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients include those who undergo uncomplicated cataract extraction surgery and IOL implantation by KLC.

Exclusion Criteria: Patients who:

1. suffer from diabetes and have more than mild background diabetic retinopathy,
2. have a history of intraocular surgery,
3. have a history of ocular trauma,
4. have known pathology of the cornea,
5. have a history of intraocular inflammation,
6. are unable to understand English,
7. are decisionally impaired,
8. are currently incarcerated, or
9. are less than 18 years of age.

No exclusions will be made on the basis of gender, ethnicity, or race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Surgically induced astigmatism | 1 month
  measured by topography at 1 month post operative visit

SECONDARY OUTCOMES:
Endothelial cell loss | one month
  As measured by specular microscopy
Best corrected visual acuity | one month
  By manifest refraction
Final incision size | intraoperatively (day #0)
  measured with incision gauges before and after lens injection.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cohen, MD, Principal Investigator — UNC dept. of ophthalmology
Locations (1):
- Kittner Eye Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Tsuneoka H, Hayama A, Takahama M. Ultrasmall-incision bimanual phacoemulsification and AcrySof SA30AL implantation through a 2.2 mm incision. J Cataract Refract Surg. 2003 Jun;29(6):1070-6. doi: 10.1016/s0886-3350(03)00076-2. PMID 12842669
- [Background] Kamae KK, Werner L, Chang W, Johnson JT, Mamalis N. Intraocular pressure changes during injection of microincision and conventional intraocular lenses through incisions smaller than 3.0 mm. J Cataract Refract Surg. 2009 Aug;35(8):1430-6. doi: 10.1016/j.jcrs.2009.03.038. PMID 19631132
- [Background] Osher RH. Microcoaxial phacoemulsification Part 2: clinical study. J Cataract Refract Surg. 2007 Mar;33(3):408-12. doi: 10.1016/j.jcrs.2006.10.055. PMID 17321390
- [Background] Kohnen T, Klaproth OK. Incision sizes before and after implantation of SN60WF intraocular lenses using the Monarch injector system with C and D cartridges. J Cataract Refract Surg. 2008 Oct;34(10):1748-53. doi: 10.1016/j.jcrs.2008.06.031. PMID 18812128
- [Background] Ventura AC, Walti R, Bohnke M. Corneal thickness and endothelial density before and after cataract surgery. Br J Ophthalmol. 2001 Jan;85(1):18-20. doi: 10.1136/bjo.85.1.18. PMID 11133705
- [Background] Masket S, Wang L, Belani S. Induced astigmatism with 2.2- and 3.0-mm coaxial phacoemulsification incisions. J Refract Surg. 2009 Jan;25(1):21-4. doi: 10.3928/1081597X-20090101-04. PMID 19244949